CLINICAL TRIAL: NCT00148837
Title: Randomized Double Blind Trial Comparing the Efficacy of Prazosin Versus Placebo Associated With Peg-Interferon Alpha 2b and Ribavirin for Initial Treatment of Patients With Hepatitis C With Genotype 1 or 4 and Severe Fibrosis
Brief Title: Efficacy of Prazosin Versus Placebo Associated With Peg-Interferon Alpha 2b and Ribavirin in Chronic Hepatitis C With Genotype 1 or 4 and Severe Fibrosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Responsible Party: Nadia Squalli/regulatory affairs, ANRS
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2004-001326-24; ANRSHC17 Prazor
Record Dates: First submitted 2005-09-07; First posted 2005-09-08 (Estimated); Last update posted 2008-02-08 (Estimated); Status verified 2008-02

CONDITIONS: Hepatitis C, Chronic; Fibrosis
Keywords: Hepatitis C, Chronic; Fibrosis; Interferon Alfa-2b; Ribavirin; Prazosin
MeSH Terms: conditions — Hepatitis C, Chronic; Fibrosis | interventions — Pharmaceutical Preparations; Ribavirin; Prazosin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Peg-interferon alpha 2b (drug)
Drug: Ribavirin (drug)
Drug: Prazosin (drug)

SUMMARY:
Viral hepatitis C prognosis is related to the presence of a fibrosis and to the risk of developing cirrhosis or hepatic cancer. The study will evaluate the efficacy of prazosin to make hepatic fibrosis regress, in patients with chronic hepatitis C and severe fibrosis.

DETAILED DESCRIPTION:
Treatment of hepatitis C with interferon and ribavirin has a virological effect. Viral hepatitis C prognosis is related to the presence of a fibrosis and to the risk of developing cirrhosis or hepatic cancer. In vitro studies of prazosin suggest an effect against hepatic fibrosis, but the clinical effect of prazosin on the hepatic fibrosis induced by hepatitis C infection is unknown. The purpose of this multicentric national study is to compare the effects among the hepatic fibrosis of peg-interferon alpha 2b and ribavirin with prazosin or not (placebo). 112 patients with a viral hepatitis C, genotype 1 or 4, and severe fibrosis, will be randomly assigned to one of two treatment groups: peg-interferon alpha 2b and ribavirin, with prazosin or with placebo. Peg-interferon alpha 2b will be administered once a week (1.5 micro g per kg) during 48 weeks, ribavirin 1,000 to 1,200 mg per day (according to weight) during 48 weeks, prazosin/placebo 5 mg (2 pills) per day during 96 weeks. Evaluation will be done at 96 weeks. The primary end-point is the proportion of patients presenting a decrease of fibrosis. Secondary end-points are other criteria of histological response, virological response, biochemical response.

ELIGIBILITY:
Inclusion Criteria:

* Chronic viral hepatitis C, genotype 1 or 4
* Fibrosis F3 or F3-F4, assessed by the scoring Metavir system
* Initial treatment against HCV

Exclusion Criteria:

* Psychiatric pathology
* Alcool consummation
* Pregnancy or plan of pregnancy
* Breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2004-09

PRIMARY OUTCOMES:
Proportion of patients presenting a decrease of fibrosis as measured on the liver biopsy and considered as clinically interesting (decrease of fibrosis pre- and post-therapeutic (W96) measures of at least 10 percent)

SECONDARY OUTCOMES:
Metavir scoring system; immunostaining of alpha-smooth muscle actin; indirect markers of fibrosis (Fibrotest) at W96
Sustained virological response: undetectable HCV RNA at W96
Sustained biochemical response: ALT level at W96

CONTACTS AND LOCATIONS:
Overall Officials: de Ledinghen Victor, MD, PhD, Principal Investigator — Hopital du Haut-Leveque, Service d'Hepato-Gastroenterologie, Pessac 33604, France; Chene Genevieve, MD, PhD, Study Director — INSERM Unite 593, Bordeaux, France
Locations (1):
- Hopital du haut Leveque, Pessac, France